CLINICAL TRIAL: NCT06603766
Title: Comparative Study Between Nebuliezed and Intravenous Magnesium Sulfate for Treatment of Persistant Pulmonary Hypertension in Neonates
Brief Title: Treatment of Persistent Pulmonary Hypertension in Neonates With Nebulized Magnesium Sulfate
Acronym: PPHN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Heba Morsy Saad El Din El Ganady, Principal investigator, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39-9-204
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Magnesium Sulfate - PPHN
Keywords: PPHN; magnesium sulfate; Neonates
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized magnesium (NebMag) group 1 (Active Comparator): NebMag group (n=20) was administered nebulized isotonic magnesium (64 mg/mL). For nebulization, an isotonic MgSO₄ solution (64 mg/mL) was formulated by diluting a 10% intravenous preparation of MgSO₄ heptahydrate with sterile distilled water. 4 mL aliquots of the isotonic MgSO₄ solution (containing 256 mg of MgSO₄) were administered every 15 minutes through the jet nebulizer connected to the ventilator during the 24 hour study period.
  Interventions: Drug: Inhalational magnesium sulfate
- Intravenous magnesium (IVMag) group 2 (Active Comparator): IVMag group (n=20) received intravenous magnesium. For intravenous administration, a 10% MgSO₄ solution was prepared by diluting a 50% intravenous formulation of MgSO₄ heptahydrate with 5% glucose and administrated in a loading dose of 2 mL/kg over 30 minutes (equivalent to 200 mg/kg of MgSO₄), followed by a continuous infusion at a rate of 0.5 mL/kg/h (equivalent to 50 mg/kg/h of MgSO₄) over the 24 hour study period.
  Interventions: Drug: IV Magnesium Sulfate

INTERVENTIONS:
Drug: IV Magnesium Sulfate — MgSO₄'s mechanism in PPHN includes activating cellular processes, modulating membrane excitability, and acting as a physiological calcium antagonist. It exerts sedative, muscle relaxant, and bronchodilatory properties, while concurrently inducing a state of alkalosis.
  Other Names: IV MgSO4
  Arms: Intravenous magnesium (IVMag) group 2
Drug: Inhalational magnesium sulfate — It gives us the same mechanism of action as IV MgSO4 with less side effects.
  Other Names: Inhalational MgSO4
  Arms: Nebulized magnesium (NebMag) group 1

SUMMARY:
we conducted this study to compare between effect of nebulized and intravenous magnesium sulfate (MgSO₄) for better treatment of persistent pulmonary hypertension of neonates with less side effects.

DETAILED DESCRIPTION:
Persistent pulmonary hypertension of the newborn (PPHN) is a serious syndrome characterized by sustained fetal elevation of pulmonary vascular resistance (PVR) at birth. The syndrome is seen in two of 1000 live-born infants and is associated with anormal or low systemic vascular resistance. Pulmonary hypertension is defined as a mean pulmonary artery pressure greater than 25 mmHg at rest and > 30 mmHg during exercise. PPHN-targeted therapy is used for infants with PPHN who fail to respond to general cardiopulmonary supportive care. Oxygen and inhaled Nitric Oxide (iNO) are the only well-studied pulmonary vasodilators in neonates with PPHN. Magnesium is a potent vasodilator and hence has the potential to reduce the high pulmonary arterial pressures as it's able to dilate constricted muscles in the pulmonary arteries. However, its action is not specific and when given via an intravenous infusion, it will act on other muscles in the body including other arteries. Excessive magnesium causes hypotonia, hypotension, and cardiorespiratory failure. However, no studies have demonstrated long-term benefit. Delivering magnesium sulfate by nebulization may enhance effectiveness and minimizes systemic adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with documented persistent pulmonary hypertension as confirmed by echocardiography.
* Neonates born at ≥ 35 wk. gestation with a birth weight of 2.5-4 kg
* Neonates have to be connected to mechanical ventilation with an oxygenation index (OI) >30 on two occasions at least 15 min apart.
* The echocardiogram had to show a predominant right-to-left or bidirectional shunt (through ductus arteriosus and/or foramen oval) and/or tricuspid regurgitant jet with a pressure gradient ≥ 2/3 of the systemic systolic blood pressure.

Exclusion Criteria:

* Infants of parents who refuse to give informed consent.
* Infants of mothers who receive magnesium sulfate within 48 h before labor.
* Congenital heart diseases other than patent ductus arteriosus (PDA) and foramen ovale.
* Major congenital anomalies, including congenital diaphragmatic hernia and lung hypoplasia.
* Prior need for cardiopulmonary resuscitation
* Mean arterial blood pressure (MABP) < 35 mmHg despite therapy with volume infusions and vasoactive inotropes.
* Impaired kidney function; and prior administration of pulmonary vasodilators or prior administration of surfactant.

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osama Z. El Feky, Professor, Study Director — Pediatrics Department, Faculty of Medicine, Benha University, Benha, Egypt.
Locations (1):
- Pediatrics Department, Faculty of Medicine, Benha University., Benha, Egypt., Egypt

IPD SHARING:
Plan to Share IPD: Undecided
demographic data, preliminary clinical data

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of neonates who admitted at Benha University hospital diagnosed as PPHN during study period was 158. 95 was excluded as they did not meet inclusion criteria. 23 parents refused to participate in the study.
Period: Overall Study
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: gestional weeks] | 37.1 (0.9) | 37.2 (1.1) | 37.15 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 11 | 10 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 20 | 20 | 40
Body weight (kg) [Mean (Standard Deviation); unit: kg] | 3.1 (0.3) | 3.1 (0.3) | 3.1 (0.3)
mode of delivery [Count of Participants; unit: Participants]
  vaginal delivery | 7 | 5 | 12
  caesarean delivery | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Airway Pressure (cm H2O)
Time Frame: from baseline to 12 and 24 hours after administering the study drug
Measure: Mean (Standard Deviation); unit: (cm H2O)
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2
Number analyzed (Participants) | 20 | 20
(cm H2O)
  Baseline | 14.1 (1.29) | 13.8 (1.18)
  At 12h | 13.7 (1) | 13.25 (0.9)
  At 24h | 14 (1.27) | 13.8 (1.24)
Statistical Analysis 1: Comparison: Nebulized Magnesium (NebMag) Group 1 vs Intravenous Magnesium (IVMag) Group 2; Test type: Superiority; p = 0.83, Chi-squared

2. Primary Outcome: Fraction of Inspired Oxygen (FiO2) (%)
Time Frame: from baseline to 12 and 24 hours after administering the study drug
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2
Number analyzed (Participants) | 20 | 20
percentage
  baseline | 100 (0) | 100 (0)
  at 12h | 96.5 (5.8) | 97.5 (4.4)
  at 24h | 96 (5.9) | 97 (5.7)
Statistical Analysis 1: Comparison: Nebulized Magnesium (NebMag) Group 1 vs Intravenous Magnesium (IVMag) Group 2; Test type: Superiority; p = 0.46, Chi-squared

3. Primary Outcome: PaO2 (mmHg)
Description: kPa x 7.5 converts to the equivalent PaO2 in mmHg
Time Frame: from baseline to 6, 12 and 24 hours after administering the study drug
Measure: Mean (Standard Deviation); unit: (mmHg)
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2
Number analyzed (Participants) | 20 | 20
(mmHg)
  Baseline | 38.45 (2) | 38.35 (1.63)
  12H | 54.8 (5.43) | 51.45 (3.46)
  24H | 69.45 (7.56) | 60.75 (5.9)
Statistical Analysis 1: Comparison: Nebulized Magnesium (NebMag) Group 1 vs Intravenous Magnesium (IVMag) Group 2; Test type: Superiority; p = 0.008, Chi-squared

4. Primary Outcome: Tracking Changes in the Oxygenation Index (OI)
Description: OI evaluates both oxygenation and ventilatory support, aiding decisions on Extracorporeal Membrane Oxygenation (ECMO) necessity in newborns with PPHN. OI calculated as (Mean Airway Pressure (cm H2O) x Fraction of Inspired Oxygen (%) x 100) ÷ (PaO2 (kPa) x 7.5).
  OI is routinely used as an indicator of severity of hypoxemic respiratory failure (HRF) in neonates, with an arbitrary cutoff of 15 or less for mild HRF, between 16 and 25 for moderate HRF, between 26 and 40 for severe HRF, and more than 40 for very severe HRF
Time Frame: from baseline to 12 and 24 hours after administering the study drug
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2
Number analyzed (Participants) | 20 | 20
index
  Baseline | 34.3 (2.4) | 34.1 (2.2)
  12h | 24.2 (2.6) | 25.1 (2.4)
  24h | 19.75 (2.9) | 22.1 (2.19)
Statistical Analysis 1: Comparison: Nebulized Magnesium (NebMag) Group 1 vs Intravenous Magnesium (IVMag) Group 2; Test type: Superiority; p = 0.032, Chi-squared

5. Secondary Outcome: the Variations in Mean Arterial Blood Pressure (MABP)
Description: Both systolic and diastolic pressure are used to calculate MABP.
Time Frame: at 0, 12, and 24 hours post administration of the study drug relative to baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2
Number analyzed (Participants) | 20 | 20
mmHg
  Baseline | 45.8 (2.7) | 45.7 (2.7)
  12h | 53.6 (3.2) | 48.6 (2.3)
  24h | 56.8 (3.3) | 53.6 (2.4)
Statistical Analysis 1: Comparison: Nebulized Magnesium (NebMag) Group 1 vs Intravenous Magnesium (IVMag) Group 2; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: the Alterations in Serum Magnesium Levels (mmol/L)
Time Frame: from baseline to 12 hours following the administration of the study drug.
Measure: Mean (Standard Deviation); unit: (mmol/L)
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2
Number analyzed (Participants) | 20 | 20
(mmol/L)
  Baseline | 0.92 (0.1) | 0.93 (0.1)
  At 12h | 1.2 (0.17) | 3.6 (0.18)
Statistical Analysis 1: Comparison: Nebulized Magnesium (NebMag) Group 1 vs Intravenous Magnesium (IVMag) Group 2; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: this study couldn't detect adverse event during 24 h study duration
Arm/Group | Nebulized Magnesium (NebMag) Group 1 | Intravenous Magnesium (IVMag) Group 2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
First, the study involved a limited group of neonates with PPHN. Second, a single dosage of magnesium was administered via continuous nebulization in this trial. It is still technically difficult to have a reliable & effective nebulization system while using mechanical breathing. Thirdly, effects of nebulized magnesium sulfate in combination with other pulmonary vasodilators were not disclosed by study. Finally, because of study's constrained time frame, critical outcomes could not be addressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT06603766/Prot_SAP_000.pdf